CLINICAL TRIAL: NCT01030367
Title: Pilot Study of Organic Nitrates on Endothelial Progenitor Cells and Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Pilot Study of Organic Nitrates on Endothelial Function in CAD Patients
Acronym: ONEEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Julius-Maximilians University (Other)
Responsible Party: Julius-Maximilians University, Julius-Maximilians University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0001
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): PETN
  Interventions: Drug: PETN, ISDN
- 2 (Experimental): ISDN
  Interventions: Drug: PETN, ISDN
- 3 (No Intervention)
  Interventions: Drug: PETN, ISDN

INTERVENTIONS:
Drug: PETN, ISDN — Oral dosing of organic nitrates PETN 2x 80mg per day ISDN 2x40mg per day

SUMMARY:
Organic nitrates increase levels of circulating endothelial progenitor cells (Thum et al., Arterioscler Thromb Vasc Biol. 2007 Apr;27(4):748-54). Here, we want to test the effects of two different organic nitrates (PETN, ISDN) on number and function of endothelial progenitor cells and endothelial function.

DETAILED DESCRIPTION:
In this pilot study we test the effects of two different organic nitrates (PETN, ISDN) on number and function of endothelial progenitor cells and endothelial function. These parameters will be measured before and after 14d of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease, 2- or 3-vessel disease

Exclusion Criteria:

* Acute myocardial infarction, acute heart failure, cancer, acute infections

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-11 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial function Number of endothelial progenitor cells Function of endothelial progenitor cells | Baseline and after 14d

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Thum, MD, PhD, Principal Investigator — University of Würzburg
Locations (1):
- Julius-Maximilians University, Würzburg, Bavaria, Germany

REFERENCES:
- [Background] Thum T, Fraccarollo D, Thum S, Schultheiss M, Daiber A, Wenzel P, Munzel T, Ertl G, Bauersachs J. Differential effects of organic nitrates on endothelial progenitor cells are determined by oxidative stress. Arterioscler Thromb Vasc Biol. 2007 Apr;27(4):748-54. doi: 10.1161/01.ATV.0000258787.18982.73. Epub 2007 Jan 25. PMID 17255540